CLINICAL TRIAL: NCT06107374
Title: Imaging of T-cell Activation With [18F]F-araG in Advanced Non-Small Cell Lung Cancer (NSCLC) Patients Undergoing PD-1/PD-L1 Directed Therapy
Brief Title: Imaging Advanced NSCLC Patients Undergoing PD-1/PD-L1 Directed Therapy Using [18F]-FARAG
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CST-FARAG-IO-UIOW-201
Record Dates: First submitted 2023-10-10; First posted 2023-10-30 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Advanced Non Small Cell Lung Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Advanced non small cell lung cancer (NSCLC) patients undergoing PD-1/PD-L1 directed therapy (Experimental)
  Interventions: Drug: [18F]F-AraG

INTERVENTIONS:
Drug: [18F]F-AraG — Two PET scans

SUMMARY:
This pilot study uses [18F]F AraG PET imaging to evaluate the immunological response to checkpoint inhibitor therapy (CkIT) in patients with advanced NSCLC tumors. The study's main objectives are to quantify the change in [18F]F AraG PET signal before and while on CkIT therapy and to correlate this change in [18F]F AraG PET signal with radiographic response.

To explore these objectives, eligible subjects will undergo pre- and on - CkIT treatment [18F]F AraG PET/CT scans, and will be followed up for 12 months for assessment of radiographic and clinical outcomes. This study is a single-site, open label, non randomized, single arm pilot trial. Patients and care providers will not be blinded to any part of the study.

DETAILED DESCRIPTION:
Checkpoint inhibitor therapy has led to impressive clinical successes, providing objective and durable responses in patients with advanced cancers that previously had few treatment options. Unfortunately, immunotherapy works only in a relatively small fraction of patients with solid tumors.

The current standard of care anatomic imaging adequately assessed treatment efficacy in the pre-immunotherapy era, when tumor volume burden directly correlated with clinical outcomes. However, anatomic imaging is found to be limited due to the cellular and molecular nature of early responses to immunotherapy. PET imaging is a sensitive technique that uses radiolabeled agents to visualize the distribution of specific molecular targets in the body. Based on its ability to pinpoint molecular activity, PET imaging agents that target key players of the immune response could offer a powerful noninvasive tool for evaluating complex immunologic processes within the body.

[18F]F-AraG was developed as an agent for imaging activated T cells. [18F]F-AraG is an 18F-labeled analog of 9-b-D-Arabinofuranosylguanine a compound that has shown selective accumulation in T cells and whose prodrug, nelarabine, is FDA-approved for the treatment of patients with T cell acute lymphoblastic leukemia and T cell lymphoblastic lymphoma. [18F]F-AraG is independent of the type of immunotherapy regimen being administered adoptive cell therapy, checkpoint inhibitors, cancer vaccines or a combination of immunotherapy and conventional medicines. In vivo, real-time imaging of activated T cells in solid tumors before and at a timepoint during and after CkIT therapy can help understand the effects of checkpoint blockade therapy. Additionally, in vivo whole-body imaging of activated T cells can provide critical information about the effect of immunomodulation in resulting in autoimmunity, and thus help predict adverse events of immunotherapy.

To sum up, characterizing the immune system alterations in vivo, in real-time, and non-invasively using PET imaging may enable us to predict better which patients will benefit from which Checkpoint Inhibitor Therapy (CkIT) treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NSCLC and planned to undergo immunotherapy as monotherapy or as combination therapy for advanced/metastatic disease.
2. Measurable disease.
3. ECOG performance status of 0, 1 or 2.
4. Subjects are willing to be followed at the University of Iowa.

Exclusion Criteria:

1. Serious comorbidities that in the opinion of the investigator/sponsor could compromise protocol objectives.
2. Pregnant women or nursing mothers.
3. Patients with severe claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
[18F]F-AraG Quantification | One Year
  Quantitative assessment of tracer uptake by Standardized Uptake Value (SUV) based measurements within volumes of interest on pre- and on-treatment [18F]F AraG PET scans compared.
[18F]F AraG Correlation | One Year
  Comparison of quantitative change in tracer uptake between pre- and on-treatment with radiographic outcomes as defined as Complete Response (CR) + Partial Response (PR) + stable disease (SD) > 4 months.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Furqan, M.D., Principal Investigator — Holden Comprehensive Cancer Center
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided